CLINICAL TRIAL: NCT04802447
Title: Expanded Access to SurVaxM for Treatment of Patients With Glioblastoma Who Have No Access to Other Comparable or Alternative Therapy or Have Completed Treatment on a Non-Randomized Clinical Trial of SurVaxM and May Benefit From Further Treatment
Brief Title: SurVaxM Expanded Access Protocol
Acronym: EAP
Status: No longer available | Type: Expanded Access
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I 546319
Record Dates: First submitted 2021-03-08; First posted 2021-03-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: SurVaxM — Each participant will receive 4 doses of SVN53-67/M57-KLH (SurVaxM) spaced two weeks apart. This phase of treatment is known as the prime-boost phase and will take 6 weeks to complete. After completion of the prime-boost phase of treatment, the participant will receive a dose ofSVN53-67/M57-KLH (SurVaxM) every 3 months for up to two years
  Other Names: SVN53-67/M57-KLH

SUMMARY:
Data from clinical trials suggest that SurVaxM administered as a single agent, or in combination with standard glioblastoma chemotherapy treatment regimens to patients with recurrent or newly diagnosed glioblastoma, is generally well tolerated and may increase progression free survival and overall survival in some patients

ELIGIBILITY:
This EAP is intended for the following patients only:

* Roswell Park patients with glioblastoma who are not eligible for an appropriate clinical trial for their glioblastoma, but who meet required eligibility criteria listed herein and,
* Roswell Park patients with glioblastoma who have completed participation in a nonrandomized clinical trial of SurVaxM, but who wish to continue to receive SurVaxM as part of their ongoing care, and who meet all other eligibility criteria listed herein and,
* Patients at institutions other than Roswell Park who have completed treatment on a nonrandomizedclinical trial of SurVaxM at their participating institution, but who wish to continue to receive SurVaxM as part of their ongoing care, and who meet all other eligibility criteria listed herein. Such patients must agree to, and be able to, participate at Roswell Park.

Inclusion Criteria:

* Patient has newly diagnosed or recurrent or progressive glioblastoma who falls under one or more exclusion criteria of another SurVaxM clinical study currently recruiting, or has completed participation in another non-randomized clinical trial of SurVaxM for glioblastoma and is off study but wishes to receive SurVaxM as part of his/her treatment
* Karnofsky performance status ≥ 70 (refer to Appendix A).
* A pathologically confirmed diagnosis of glioblastoma of the brain or spinal cord is required, unless biopsy is determined by the PI not to be in the patient's best interest.
* Have the following clinical laboratory values obtained within 28 days prior to registration:
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* Creatinine ≤ 1.8 mg/dL
* Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin or oral anticoagulants) must meet the following criteria:
* No active bleeding or pathological condition that carries a high risk of bleeding (e.g., coagulopathy)
* For participants of child-bearing potential: must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to enrollment and, have a negative pregnancy test prior to starting treatment under this protocol.
* Dose of corticosteroids reduced to the minimum required to control neurologic symptoms.
* Patients with newly diagnosed glioblastoma must have completed radiation therapy and temozolomide or "standard of care" treatment of their glioblastoma, unless it is determined by their treating physician that it is not in the best interest of the patient to do so.
* Participant must understand the investigational nature of this study drug and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving SurVaxM.
* Patient is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.

Exclusion Criteria:

* Patient meets all inclusion criteria for another SurVaxM clinical study that is open and recruiting.
* Patient has previously participated in a clinical trial in which randomization to an arm with SurVaxM treatment was part of the trial design..
* Patients with newly diagnosed or recurrent glioblastoma who have not had standard of care treatment with fractionated radiation therapy and temozolomide, unless these treatments have been determined to be medically contraindicated or are not tolerate.
* Patient's brain tumor has not been biopsied, unless biopsy is determined by the PI not to be in the patient's best interest.
* Patient has serious concurrent infection or medical illness, which in the treating physician's opinion would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* History of tuberculosis, granulomatous disease or systemic autoimmune disorder.
* Patient is pregnant or breast-feeding.
* Concurrent participation in any clinical therapeutic studies involving investigational drug(s) (Phases 1-4).
* Patient has concurrent or prior malignancy except curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for at least 2 years may be eligible for treatment under this protocol.
* Patient who is receiving any other concurrent chemotherapeutic agents or investigational drugs.
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness.
* Patient is unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion makes the candidate unsuitable to receive the study drug or protocol procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Abad, MD, Principal Investigator — Roswell Park Cancer Institute